CLINICAL TRIAL: NCT07350590
Title: Short- and Long-Term Outcomes of Robotic vs. Laparoscopic Right Hemicolectomy: A Multicenter Retrospective Study
Brief Title: Comparison Between Robotic and Laparoscopic Right Hemicolectomy
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Principal Investigator, Sir Run Run Shaw Hospital
Other Study IDs: LRCRC
Record Dates: First submitted 2026-01-03; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Right-sided Colon Cancer
Keywords: right-sided colon cancer; robotic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic right hemicolectomy
  Interventions: Procedure: laparoscopic right hemicolectomy
- robotic right hemicolectomy
  Interventions: Procedure: robotic right hemicolectomy

INTERVENTIONS:
Procedure: laparoscopic right hemicolectomy — laparoscopic right hemicolectomy
  Groups: laparoscopic right hemicolectomy
Procedure: robotic right hemicolectomy — robotic right hemicolectomy
  Groups: robotic right hemicolectomy

SUMMARY:
This study aims to compare outcomes of robotic versus laparoscopic right hemicolectomy for right colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* colon cancer lesions to be located at the hepatic flexure, ascending colon, or cecum, as confirmed by colonoscopy
* the pathological biopsy revealed adenocarcinoma, and the clinical staging was diagnosed as clinical stages I to IV according to the American Joint Committee on Cancer (AJCC) TNM classification (8th edition)
* the patients plan to undergo right hemicolectomy
* the Eastern Cooperative Oncology Group Performance Status (ECOG-PS) is 0 or 1

Exclusion Criteria:

* incomplete case data
* surgery performed after colorectal cancer recurrence
* patients with multiple primary cancers and other malignant tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: right colon cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Disease free survival(DFS) | 3 years after surgery
  The three-year disease-free survival of patients.

SECONDARY OUTCOMES:
Overall survival(OS） | 3 years after surgery
  The three-year overall survival of patients.
Surgical complications | During the perioperative period
  During the perioperative period, the incidence of surgical complications
Surgical recovery time | During the perioperative period
  It refers to the time required for patients to resume gas passing, bowel movements, be discharged from the hospital, and return to normal life after surgery
Hospitalization expenses | During the perioperative period
  Hospitalization expenses include surgery-related costs

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided